CLINICAL TRIAL: NCT01140893
Title: Effects of EXEnatide on Glycemic Control and Weight Over 26 Weeks in Continuous Subcutaneous Insulin Infusion (CSII) Treated Patients With Type 2 Diabetes : a Phase 2/3 Double Blind randoMized Placebo-controlled Trial.
Brief Title: Effects of Exenatide on Glycemic Control and Weight in Continuous Subcutaneous Insulin Infusion (CSII) Type 2 Treated Patients With Type 2 Diabetes
Acronym: EXEPUMP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT N° 2009-016384-11
Record Dates: First submitted 2010-05-03; First posted 2010-06-10 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; CSII; Exenatide; Double Blind Placebo Controlled Study
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exenatide (Experimental): 55 subjects
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): 55 subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Research drug (exenatide or placebo), will begin at V0, after randomization. The initial dosage for the first month will be 5 µg SC BID. Injections can be administered at any time within the 60 minute period before the morning and evening meal.
  From V1, research drug will be titrated from 5 to 10 µg SC BID. If gastro-intestinal adverse effects occur with 10 µg SC BID, the dosage will be back-titrated to 5 µg SC BID. Thus, the higher research drug dosage tolerated will be used during the study time.
  Other Names: Exenatide = BYETTA (R)
  Arms: exenatide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether exenatide is effective to improve glycemic control among type 2 diabetic patients treated by insulin pump therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 35 to 70
* Type 2 diabetes diagnosed for at least 12 months, according the criteria of the American Diabetes Association :

  * presence of classic symptoms of diabetes mellitus with unequivocal elevation of plasma glucose (2-hour post-prandial or random glucose >200 mg/dL) or
  * fasting plasma glucose elevation on more than 1 occasion > 125 mg/dL or
  * patient currently undergoing pharmacological and/or non-pharmacological treatment for diabetes mellitus
* CSII treatment using a rapid analog for at least 6 month (CSII being initiated in patients with HbA1c > 8 % despite a well-conducted MDI trial using a 2 to 5 daily injection regimen)
* HbA1c ≥ 7,5% and ≤ 10 %
* BMI ≥ 25 and ≤ 45
* Stable body weight (≤10% variation) during the 3 last months

Exclusion Criteria:

* Type 1 diabetes assessed by positive anti-GAD65 or anti-insulin or anti-IA2 antibodies
* Monogenic diabetes (MODY, mitochondrial diabetes…)
* Current treatment with OHA (OHA ought to be interrupted at least two months prior to inclusion in the study)
* Current treatment specifically addressed for weight lost (orlistat, sibutramine, rimonabant may be interrupted at least 3 months prior to inclusion in the study)
* Use of corticosteroid therapy for more than 10 days within the 3-past months, or patient who ought to be treated by corticosteroid during the study period
* Clinically significant hepatic disease
* Documented gastroparesis, or current use of drugs that directly affect gastrointestinal motility, or any significant abdominal disease that may increase the risk of adverse gastrointestinal effects induced by exenatide
* Kidney failure (MDRD less than 50 ml/min)
* Pregnancy/breastfeeding
* Any social and/or mental condition rendering the subject unable to understand the scope and possible consequences of the study
* Concurrent enrolment in another clinical trial
* Geographically inaccessible for follow-up visits required by protocol

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-11; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 6 months of centrally measured HbA1c | baseline to 6 months

SECONDARY OUTCOMES:
Change from baseline in weight, BMI, waist circumference, 6 points glucose profile, insulin doses, % of daily use of insulin as basal rate, % of daily use of insulin as bolus, quality of life questionnaire | baseline to 6 months
Change from baseline in mean blood glucose value | baseline to 6 months
  occurrence of hyperglycemia above 190 mg/dl expressed as Area under the Curve (high) above 190 mg/dl (10.5 mmol/l), occurrence of hypoglycemia below 70 mg/dl (3.9 mmol/l) expressed as Area Under the Curve (low) below 70 mg/dl, glycemic variability (MAGE index).

CONTACTS AND LOCATIONS:
Overall Officials: Michael JOUBERT, MD, Principal Investigator — Endocrinology Unit, University Hospital of Caen, FRANCE; Yves REZNIK, MD, Principal Investigator — Endocrinology Unit, University Hospital of Caen, FRANCE
Locations (3):
- France (3):
  - Endocrinology Unit and Clinical Research Center Basse Normandie, University Hospital of Caen, Caen
  - CERIDT, Corbeil-Essonne
  - Endocrinology Unit, Strasbourg